CLINICAL TRIAL: NCT04203693
Title: Observational Study to Assess the Effectiveness, Safety Profile and Real-life Prescribing and Utilization Patterns of Tildrakizumab (Ilumetri®) in Patients With Moderate to Severe Plaque Psoriasis in Routine Clinical Practice. (SAIL)
Brief Title: Observational Study of Tildrakizumab in Patients With Moderate to Severe Plaque Psoriasis in Routine Clinical Practice
Acronym: SAIL
Status: Completed | Type: Observational
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS Study M-14745-43
Record Dates: First submitted 2019-12-10; First posted 2019-12-18 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Plaque Psoriasis
Keywords: Ilumetri®; Tildrakizumab; Moderate to severe plaque psoriasis
MeSH Terms: interventions — tildrakizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: Tildrakizumab Treated Participants: Participants will be treated with tildrakizumab who have participated in prior tildrakizumab studies
  Interventions: Drug: Tildrakizumab
- Cohort 2: Newly Tildrakizumab Prescribed Participants: Participants will be newly prescribed tildrakizumab (a prescription has occurred independently of the enrolment in the study)
  Interventions: Drug: Tildrakizumab

INTERVENTIONS:
Drug: Tildrakizumab — The study physicians will choose the treatment independently of the enrolment in the study according to routine care.

SUMMARY:
The observational, non-interventional study will assess the efficacy, safety, prescription and utilization patterns of Tildrakizumab in participants with moderate to severe plaque psoriasis in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent form.
* Age >= 18years.
* Moderate to severe chronic plaque psoriasis diagnosis.
* Participants who have participated in Tildrakizumab (Ilumetri®) clinical trials (Cohort 1) OR participants who, according to the physician's therapeutic decision, should start the treatment with Tildrakizumab (Ilumetri®) (Cohort 2).

Exclusion Criteria:

* Unable to comply with the requirements of the study or who in the opinion of the study physician should not participate in the study.
* Participants meeting any of the exclusion criteria specified in the summary of product characteristics (SmPC) of Ilumetri®.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female patients with moderate-to-severe chronic plaque psoriasis.
Sampling Method: Non-Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Cohort 1: Absolute Psoriasis Area and Severity Index (PASI) at Week 48 | Week 48
  PASI is a combined assessment of lesion severity and affected area into a single score.
Cohort 1: Absolute Psoriasis Area and Severity Index (PASI) at Week 96 | Week 96
  PASI is a combined assessment of lesion severity and affected area into a single score.
Cohort 1: Change From Baseline in Psoriasis Area and Severity Index at Week 48 | Baseline (Day 0) and Week 48
  PASI is a combined assessment of lesion severity and affected area into a single score.
Cohort 1: Change From Baseline in Psoriasis Area and Severity Index at Week 96 | Baseline (Day 0) and Week 96
  PASI is a combined assessment of lesion severity and affected area into a single score.
Cohort 1: Correlation Between Absolute Psoriasis Area and Severity Index Scores and Dermatology Life Quality Index adjusted for not relevant responses (DLQI-R) at Week 48 | Week 48
  PASI is used to assess the lesion severity and affected area due to psoriasis. Dermatology Life Quality Index (DLQI) questionnaire is the most commonly used tool to assess the effect of skin diseases on a subject's quality of life. Dermatology Life Quality Index adjusted for not relevant responses (DLQI-R) is a newly introduced variation of the regular DLQI that adjusts the total score for the number of not relevant responses.
Cohort 1: Correlation Between Absolute Psoriasis Area and Severity Index Scores and Dermatology Life Quality Index adjusted for not relevant responses (DLQI-R) at Week 96 | Week 96
  PASI is used to assess the lesion severity and affected area due to psoriasis. Dermatology Life Quality Index (DLQI) questionnaire is the most commonly used tool to assess the effect of skin diseases on a subject's quality of life. Dermatology Life Quality Index adjusted for not relevant responses (DLQI-R) is a newly introduced variation of the regular DLQI that adjusts the total score for the number of not relevant responses.
Cohort 1: Percentage of Participants who maintaining Psoriasis Area and Severity Index 75, 90, and 100 Responses at Week 48 | Week 48
  PASI is a combined assessment of lesion severity and affected area into a single score.
Cohort 1: Percentage of Participants who maintaining Psoriasis Area and Severity Index 75, 90, and 100 Responses at Week 96 | Week 96
  PASI is a combined assessment of lesion severity and affected area into a single score.
Cohort 1: Absolute Body Surface Area Affected by Psoriasis (BSA) at Week 48 | Week 48
  BSA is a numerical score used to measure the total area of the body affected by psoriasis.
Cohort 1: Absolute Body Surface Area Affected by Psoriasis (BSA) at Week 96 | Week 96
  BSA is a numerical score used to measure the total area of the body affected by psoriasis.
Cohort 1: Change from Baseline in Body Surface Area Affected by Psoriasis at Week 48 | Baseline (Day 0) and Week 48
  BSA is a numerical score used to measure the total area of the body affected by psoriasis.
Cohort 1: Change from Baseline in Body Surface Area Affected by Psoriasis at Week 96 | Baseline (Day 0) and Week 96
  BSA is a numerical score used to measure the total area of the body affected by psoriasis.
Cohort 1: Absolute Physician's Global Assessment (PGA) (General, Nail, Scalp) Scores at Week 48 | Week 48
  PGA is a 5-point measure of psoriasis based on the degree of erythema, induration, and scale averaged over the entire body.
Cohort 1: Absolute Physician's Global Assessment (PGA) (General, Nail, Scalp) Scores at Week 96 | Week 96
  PGA is a 5-point measure of psoriasis based on the degree of erythema, induration, and scale averaged over the entire body.
Cohort 1: Change From Baseline in Physician's Global Assessment (PGA) (General, Nail, Scalp) at Week 48 | Baseline (Day 0) and Week 48
  PGA is a 5-point measure of psoriasis based on the degree of erythema, induration, and scale averaged over the entire body. PGA of psoriasis in general, at nail and scalp will be graded from 0 (none/clear) to 4 (severe).
Cohort 1: Change From Baseline in Physician's Global Assessment (PGA) (General, Nail, Scalp) at Week 96 | Baseline (Day 0) and Week 96
  PGA is a 5-point measure of psoriasis based on the degree of erythema, induration, and scale averaged over the entire body. PGA of psoriasis in general, at nail and scalp will be graded from 0 (none/clear) to 4 (severe).
Cohort 2: Absolute Psoriasis Area and Severity Index (PASI) at Week 52 | Week 52
  PASI is a combined assessment of lesion severity and affected area into a single score.
Cohort 2: Absolute Psoriasis Area and Severity Index (PASI) at Week 100 | Week 100
  PASI is a combined assessment of lesion severity and affected area into a single score.
Cohort 2: Change From Baseline in Psoriasis Area and Severity Index at Week 52 | Baseline (Week 0) and Week 52
  PASI is a combined assessment of lesion severity and affected area into a single score.
Cohort 2: Change From Baseline in Psoriasis Area and Severity Index at Week 100 | Baseline (Week 0) and Week 100
  PASI is a combined assessment of lesion severity and affected area into a single score.
Cohort 2: Correlation between absolute Psoriasis Area and Severity Index scores and Dermatology Life Quality Index adjusted for not relevant responses at Week 52 | Week 52
  PASI is used to assess the lesion severity and affected area due to psoriasis. Dermatology Life Quality Index (DLQI) questionnaire is the most commonly used tool to assess the effect of skin diseases on a subject's quality of life. Dermatology Life Quality Index adjusted for not relevant responses (DLQI-R) is a newly introduced variation of the regular DLQI that adjusts the total score for the number of not relevant responses.
Cohort 2: Correlation between absolute Psoriasis Area and Severity Index scores and Dermatology Life Quality Index adjusted for not relevant responses at Week 100 | Week 100
  PASI is used to assess the lesion severity and affected area due to psoriasis. Dermatology Life Quality Index (DLQI) questionnaire is the most commonly used tool to assess the effect of skin diseases on a subject's quality of life. Dermatology Life Quality Index adjusted for not relevant responses (DLQI-R) is a newly introduced variation of the regular DLQI that adjusts the total score for the number of not relevant responses.
Cohort 2: Percentage of Participants who Achieved Psoriasis Area and Severity Index 75, 90, and 100 Responses at Week 52 | Week 52
  PASI is a combined assessment of lesion severity and affected area into a single score.
Cohort 2: Percentage of Participants who Achieved Psoriasis Area and Severity Index 75, 90, and 100 Responses at Week 100 | Week 100
  PASI is a combined assessment of lesion severity and affected area into a single score.
Cohort 2: Absolute Body Surface Area Affected by Psoriasis (BSA) at Week 52 | Week 52
  BSA is a numerical score used to measure the total area of the body affected by psoriasis.
Cohort 2: Absolute Body Surface Area Affected by Psoriasis (BSA) at Week 100 | Week 100
  BSA is a numerical score used to measure the total area of the body affected by psoriasis.
Cohort 2: Change from Baseline in Percent Body Surface Area Affected by Psoriasis (BSA) at Week 52 | Baseline and Week 52
  BSA is a numerical score used to measure the total area of the body affected by psoriasis.
Cohort 2: Change from Baseline in Percent Body Surface Area Affected by Psoriasis (BSA) at Week 100 | Baseline and Week 100
  BSA is a numerical score used to measure the total area of the body affected by psoriasis.
Cohort 2: Absolute Physician's Global Assessment (PGA) (General, Nail and Scalp) at Week 52 | Week 52
  PGA is a 5-point measure of psoriasis based on the degree of erythema, induration, and scale averaged over the entire body.
Cohort 2: Absolute Physician's Global Assessment (PGA) (General, Nail and Scalp) at Week 100 | Week 100
  PGA is a 5-point measure of psoriasis based on the degree of erythema, induration, and scale averaged over the entire body.
Cohort 2: Change From Baseline in Physician's Global Assessment (PGA) (Scores of General, Nail and Scalp) at Week 52 | Baseline (Day 0) and Week 52
  PGA is a 5-point measure of psoriasis based on the degree of erythema, induration, and scale averaged over the entire body.
Cohort 2: Change From Baseline in Physician's Global Assessment (PGA) (Scores of General, Nail and Scalp) at Week 100 | Baseline (Day 0) and Week 100
  PGA is a 5-point measure of psoriasis based on the degree of erythema, induration, and scale averaged over the entire body.

SECONDARY OUTCOMES:
Absolute Dermatology Life Quality Index and Dermatology Life Quality Index Adjusted for not Relevant Responses at Week 48 and Week 96 for Cohort 1 and Week 52 and Week 100 for Cohort 2 | Cohort 1: Week 48 and Week 96; Cohort 2: Week 52 and Week 100
  Dermatology Life Quality Index (DLQI) questionnaire is the most commonly used tool to assess the effect of skin diseases on a subject's quality of life. Dermatology Life Quality Index adjusted for not relevant responses (DLQI-R) is a newly introduced variation of the regular DLQI that adjusts the total score for the number of not relevant responses.
Change from Baseline in Absolute Dermatology Life Quality Index and Dermatology Life Quality Index Adjusted for not Relevant Responses at Week 48 and Week 96 for Cohort 1 and Week 52 and Week 100 for Cohort 2 | Cohort 1: Baseline (Day 0), Week 48 and Week 96; Cohort 2: Baseline, Week 52 and Week 100
  Dermatology Life Quality Index (DLQI) questionnaire is the most commonly used tool to assess the effect of skin diseases on a subject's quality of life. Dermatology Life Quality Index adjusted for not relevant responses (DLQI-R) is a newly introduced variation of the regular DLQI that adjusts the total score for the number of not relevant responses.
Itch and Pain Visual Analogue Scales (VAS) Scores | Baseline (Day 0) to Week 96/100
  Itch and pain of the skin will be assessed by the participant on visual analogue scales (VAS).
Change from Baseline in Itch and Pain Visual Analogue Scales Scores | Baseline (Day 0) to Week 96/100
  Itch and pain of the skin will be assessed by the participant on visual analogue scales (VAS).
Number of participants who Used Concomitant Medications From Baseline at Week 48 and 96 for Cohort 1 and Week 52 and 100 for Cohort 2 | Cohort 1: Baseline (Day 0), Week 48 and Week 96; Cohort 2: Baseline, Week 52 and Week 100
  Concomitant topical, photo- or systemic anti-psoriatic and non-psoriasis therapy will be assessed.
Change from Baseline in Body Weight at End of study (EOS)/End of treatment (ET) | Baseline (Day 0) and Week 96/100 (EOS)/ET
  Change in the body weight measurement will be assessed.
Change from Baseline in Waist and hip Circumference at EOS/ET | Baseline (Day 0) and Week 96/100 (EOS)/ET
  Change in waist and hip circumference will be assessed.
Change from Baseline in Body Mass Index (BMI) at EOS/ET | Baseline (Day 0) and Week 96/100 (EOS)/ET
  Change in BMI will be assessed.
Change from Baseline in Blood Pressure at EOS/ET | Baseline (Day 0) and Week 96/100 (EOS)/ET
  Change in Blood Pressure will be assessed.
Change from Baseline in Food Intake up to EOS/ET | Baseline (Day 0) to Week 96/100 (EOS)/ET
  Participants will be asked to complete a simple questionnaire regarding their food intake.
Change from Baseline in Physical Activity up to EOS/ET | Baseline (Day 0) to Week 96/100 (EOS)/ET
  Participants will be asked to complete a simple questionnaire regarding their physical activity.
Change from baseline in Lipid Profiles up to EOS | Baseline (Day 0) to Week 96/100 (EOS)
  Serum lipid will be assessed, if available
Number of Participants Withdraw From the Study Overtime | Baseline (Day 0) to Week 96/100 (EOS)
  Participants who discontinue treatment prior to the regular end of the observation period.
Number of Participants who Underwent Dose Change up to EOS/ET | Baseline (Day 0) to Week 96/100 (EOS)/ET
  The number of participants who underwent dose change (100 mg or 200 mg).
Drug Survival up to EOS/ET | Baseline (Day 0) to Week 96/100 (EOS)/ET
  Drug survival is defined as the time from initiation of therapy to discontinuation.
Number of Participant's With Adherence to Treatment up to EOS/ET | Baseline (Day 0) to Week 96/100 (EOS)/ET
  Number of Participant's who adhere to the treatment will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Almirall, S.A.
Locations (22):
- Investigator Site 1, Vienna, Austria
- Germany (13):
  - Investigational site 5, Augsburg
  - Investigational site 10, Berlin
  - Investigational site 11, Berlin
  - Investigational site 13, Berlin
  - Investigational site 8, Erlangen
  - Investigational site 9, Greifswald
  - Investigational site 1, Hamburg
  - Investigational site 2, Hamburg
  - Investigational site 7, Kiel
  - Investigational site 3, Lübeck
  - Investigational site 6, München
  - Investigational site 12, Oberursel
  - Investigational site 4, Quedlinburg
- Italy (7):
  - Investigational site 6, Catania
  - Investigational site 7, Genova
  - Investigational site 3, Modena
  - Investigational site 4, Parma
  - Investigational site 1, Roma
  - Investigational site 2, Roma
  - Investigational site 5, Roma
- Investigational site 1, Breda, Netherlands